CLINICAL TRIAL: NCT01305642
Title: Individualized Fortification of Breast Milk for Preterm Infants - A Pilot Study
Acronym: IFO Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Christoph Fusch, Professor and Division Head, McMaster Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201101IFOPILOT
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Postnatal Growth Disorder
Keywords: Postnatal development; Breast milk fortification; Composition of breast milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individualized fortification of breast milk (Experimental)
  Interventions: Dietary Supplement: Individualized fortification of breast milk

INTERVENTIONS:
Dietary Supplement: Individualized fortification of breast milk — Lactose, fat and protein content will be measured prior to breast milk fortification.
  Subsequently, breast milk for preterm infants will individually fortified adjusted by using data from milk analysis.

SUMMARY:
To analyze the weight gain of very low birth weight infants during a minimum period of three weeks before 36 weeks postmenstrual age when infants are fed with breast milk that has been individually fortified.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≤ 1500g and gestational age < 32weeks
* Tolerating an enteral intake of ≥ 100 ml/kg/d for ≥ 24h

Exclusion Criteria:

* Infants fed more than 25% of mean caloric intake for a consecutive week with formula milk
* gastrointestinal malformation, major congenital anomalies and chromosomal abnormalities
* Babies with enterostoma or short gut syndrome
* Fluid restriction below
* Renal disease
* Sepsis
* Necrotizing enterocolitis
* Hepatic dysfunction

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
growth | from inclusion at postmentrual age <32 weeks until 36 weeks
  weight gain will be accessed three times per week

SECONDARY OUTCOMES:
enteral energy intake | from inclusion at postmentrual age <32 weeks until 36 weeks
  caloric intake by enteral feeding will be assesed daily
growth, tolerance, morbidity | from inclusion at postmentrual age <32 weeks until 36 weeks
  gains in length and head circumference will be assessed weekly, tolerance and morbidity throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Fusch, MD,PhD,FRCPC, Principal Investigator — McMaster Children's Hospital
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Fusch G, Choi A, Rochow N, Fusch C. Quantification of lactose content in human and cow's milk using UPLC-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Dec 1;879(31):3759-62. doi: 10.1016/j.jchromb.2011.09.053. Epub 2011 Oct 6. PMID 22041090
- [Background] Fusch G, Rochow N, Choi A, Fusch S, Poeschl S, Ubah AO, Lee SY, Raja P, Fusch C. Rapid measurement of macronutrients in breast milk: How reliable are infrared milk analyzers? Clin Nutr. 2015 Jun;34(3):465-76. doi: 10.1016/j.clnu.2014.05.005. Epub 2014 May 17. PMID 24912866
- [Background] Fusch G, Mitra S, Rochow N, Fusch C. Target fortification of breast milk: levels of fat, protein or lactose are not related. Acta Paediatr. 2015 Jan;104(1):38-42. doi: 10.1111/apa.12804. Epub 2014 Oct 2. PMID 25213193
- [Background] Rochow N, Landau-Crangle E, Fusch C. Challenges in breast milk fortification for preterm infants. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):276-84. doi: 10.1097/MCO.0000000000000167. PMID 25807355
- [Background] Rochow N, Fusch G, Zapanta B, Ali A, Barui S, Fusch C. Target fortification of breast milk: how often should milk analysis be done? Nutrients. 2015 Apr 1;7(4):2297-310. doi: 10.3390/nu7042297. PMID 25835073
- [Background] Fusch G, Kwan C, Huang RC, Rochow N, Fusch C. Need of quality control programme when using near-infrared human milk analyzers. Acta Paediatr. 2016 Mar;105(3):324-5. doi: 10.1111/apa.13305. Epub 2016 Jan 19. No abstract available. PMID 26663457
- [Background] Choi A, Fusch G, Rochow N, Fusch C. Target Fortification of Breast Milk: Predicting the Final Osmolality of the Feeds. PLoS One. 2016 Feb 10;11(2):e0148941. doi: 10.1371/journal.pone.0148941. eCollection 2016. PMID 26863130
- [Background] Kotrri G, Fusch G, Kwan C, Choi D, Choi A, Al Kafi N, Rochow N, Fusch C. Validation of Correction Algorithms for Near-IR Analysis of Human Milk in an Independent Sample Set-Effect of Pasteurization. Nutrients. 2016 Feb 26;8(3):119. doi: 10.3390/nu8030119. PMID 26927169
- [Result] Rochow N, Fusch G, Choi A, Chessell L, Elliott L, McDonald K, Kuiper E, Purcha M, Turner S, Chan E, Xia MY, Fusch C. Target fortification of breast milk with fat, protein, and carbohydrates for preterm infants. J Pediatr. 2013 Oct;163(4):1001-7. doi: 10.1016/j.jpeds.2013.04.052. Epub 2013 Jun 12. PMID 23769498